CLINICAL TRIAL: NCT00002200
Title: A 1592U89 Open-Label Protocol for Adult Patients With HIV-1 Infection.
Brief Title: A Study of 1592U89 in HIV-Infected Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 238M; CNAA3008
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-12

CONDITIONS: HIV Infections
Keywords: HIV-1; Administration, Oral; CD4 Lymphocyte Count; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; abacavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir

INTERVENTIONS:
Drug: Abacavir sulfate

SUMMARY:
The purpose of this study is to see if it is safe and effective to give 1592U89 to HIV-positive adults. This study also examines the influence previous anti-HIV treatment has on the effectiveness of 1592U89.

DETAILED DESCRIPTION:
Patients receive open-label 1592U89 administered orally in combination with at least one other antiretroviral agent that the patient has not previously received.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Erythropoietin, G-CSF and GM-CSF.

Patients must have:

* CD4+ cell count < 100 cells/mm3.
* HIV-1 RNA > 30,000 copies/ml.
* Signed, informed consent from parent or legal guardian for patient under 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Renal failure requiring dialysis.
* Hepatic failure evident by grade 3/4 hyperbilirubinemia and AST 5 times the upper limit of normal.
* Documented hypersensitivity to 1592U89.
* Serious medical conditions, such as diabetes, congestive heart failure, cardiomyopathy, or other cardiac dysfunction, that would compromise the safety of the patient.
* Participation in or ability to participate in an enrolling study of 1592U89.

Required:

At least 2 nucleoside reverse transcriptase inhibitors (NRTI) and one protease inhibitor (or intolerance to one protease inhibitor and one NRTI due to trying at least 2 different regimens with at least one protease inhibitor).

Alcohol or illicit drug use that may interfere with the patient's compliance.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States